CLINICAL TRIAL: NCT03718494
Title: Prevention of Alzheimer's Disease in Women: Risks and Benefits of Hormone Therapy -Continuation of: "The Kronos Early Estrogen Prevention Study (KEEPS)"
Brief Title: Continuation of The Kronos Early Estrogen Prevention Study (KEEPS)
Acronym: KEEPS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Columbia University (Other); Yale University (Other); Utah State University (Other); Brigham and Women's Hospital (Other); Banner Alzheimer's Institute (Other); University of California, San Francisco (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kejal Kantarci, Professor of Radiology, Cons-Research Neuroradiology, Mayo Clinic
Other Study IDs: 12-008697; 1RF1AG057547-01 (NIH)
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — Diagnostic Imaging; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Menopausal Hormone Therapy (mHT) Group: Women that participated in and completed the KEEPS study (NCT00154180) that were randomized to receive menopausal hormone therapy (mHT) will have a follow up brain Positron Emission Tomography (PET) imaging (F-18 Florbetapir PET or F-18 AV-1451 PET) and cognitive function testing.
  Interventions: Diagnostic Test: Brain Magnetic Resonance Imaging (MRI); Diagnostic Test: F-18 Florbetapir Positron Emission Tomography (PET) Imaging; Diagnostic Test: F-18 AV-1451 Positron Emission Tomography (PET) Imaging; Other: Neuropsychological Testing
- Placebo Group: Women that participated in and completed the KEEPS study (NCT00154180) that were randomized to receive placebo treatment will have a follow up brain Positron Emission Tomography (PET) imaging (F-18 Florbetapir PET or F-18 AV-1451 PET) and cognitive function testing.
  Interventions: Diagnostic Test: Brain Magnetic Resonance Imaging (MRI); Diagnostic Test: F-18 Florbetapir Positron Emission Tomography (PET) Imaging; Diagnostic Test: F-18 AV-1451 Positron Emission Tomography (PET) Imaging; Other: Neuropsychological Testing

INTERVENTIONS:
Diagnostic Test: Brain Magnetic Resonance Imaging (MRI) — Performed on a single 3T system and sequences will be acquired in a single sitting with an exam time under 45 minutes.
Diagnostic Test: F-18 Florbetapir Positron Emission Tomography (PET) Imaging — After a 50-minute uptake period, the patient will be positioned on the scanner bed with instructions to remain motionless. Injection of 10 mCi of 18F-Florbetapir (target dose 370 MBq, range 296 - 444 MBq) given. A helical CT image will be obtained at 50 minutes after injection of 18F-Florbetapir, followed by a 20-minute PET acquisition consisting of four 5-minute dynamic frames.
Diagnostic Test: F-18 AV-1451 Positron Emission Tomography (PET) Imaging — Intravenous bolus injection of approximately 370 MBq (10 mCi) of 18F- AV-1451 (approved under IND 124449). PET/CT image acquisition will include a low dose CT and then a 20-minute PET acquisition starting at 50-60 minutes after injection of 18F-T807 and will be performed as 4, 5-minute frames that will then be summed into one static frame. Serial frames will allow for adjustment in the case of patient motion.
Other: Neuropsychological Testing — A comprehensive battery of standardized neuropsychological tests administered by trained personnel.

SUMMARY:
The purpose of this study is to investigate how blood flow to the brain affects cognition in women who are postmenopausal, and how the use of hormone therapy early in menopause might change brain function. The testing in this study will add to the knowledge about brain aging in women. Researchers will determine if blood flow to the brain, brain structure, and cognition differences among women who took hormones in the past as part of Kronos Early Estrogen Prevention Study (KEEPS; NCT00154180), are currently taking hormones, or never took menopausal hormones.

DETAILED DESCRIPTION:
This is a continuation of the Kronos Early Estrogen Prevention Study (KEEPS) (KEEPS; NCT00154180), a multicenter double blinded, placebo-controlled, randomized trial funded by the Kronos Longevity Research Institute, Phoenix, AZ to test the hypothesis that hormone therapy started early in menopause (within the "window of opportunity") would slow progression of atherosclerosis as measured by changes in carotid artery intima-medial thickening and coronary arterial calcification.

This study will involve a single follow-up evaluation of brain imaging and cognitive function of women who were randomized to menopausal hormone therapy (mHT) or placebo, approximately 13 years post-randomization and nine years after the end of mHT administration phase in KEEPS (NCT00154180). No interventions are given as part of this study; any current hormonal treatments are by choice and prescribed by the participant's personal physician.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the original KEEPS trial.
* Able to understand study procedures.
* Willing to sign an authorization of consent in order to participate in this study.

Exclusion Criteria:

• Women who have contraindications to MRI or PET for safety reasons, such as an MRI-incompatible implant or claustrophobia.

Ages: 49 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women that participated in the Kronos Early Estrogen Prevention Study (KEEP; NCT00154180) and completed brain imaging or cognitive testing and indicated that it would be acceptable to contact them for future research opportunities.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Aβ PET SUVR | 4 years
  This measure is derived from a PET imaging study that images the deposition of the amyloid plaques of Alzheimer's disease in the brain
WMH volume | 4 years
  This measure is derived from an MRI study that images the brain structure. WMH is measured from specific regions of the brain that are vulnerable to cerebrovascular disease related injury.
Regional cortical thickness | 4 years
  This measure is derived from an MRI study that images the brain structure. The cortical thickness is measured from specific regions of the brain that are vulnerable to Alzheimer's disease related neurodegeneration.
AV-1451 | 4 years
  This measure is derived from a PET imaging study that images the deposition of the tau protein of Alzheimer's disease in the brain
Global cognitive function | 4 years
  This measurement is derived from multiple neuropsychometric tests that measure various cognitive abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Kejal Kantarci, M.D., Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Banner Health, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Study data will be de-identified and transferred to the Mayo Clinic and UW through secure file transfer protocols. Data will be stored at each institution's data center.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03718494/Prot_SAP_000.pdf